CLINICAL TRIAL: NCT07353294
Title: A Phase Ib Prospective Clinical Study Evaluating the Safety and Efficacy of Propranolol Combined With Tislelizumab Plus Gemcitabine/Cisplatin as Neoadjuvant Therapy for cT1-4aN1-3M0 Bladder Urothelial Carcinoma
Brief Title: Propranolol With Tislelizumab Plus GC in Neoadjuvant Bladder UC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2025-837-02
Record Dates: First submitted 2025-12-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Bladder Urothelial Carcinoma; Lymph Node Metastasis
Keywords: Bladder urothelial carcinoma; Lymph Node Metastasis; Neoadjuvant therapy; Tislelizumab; Gemcitabine; Cisplatin; Propranolol
MeSH Terms: conditions — Lymphatic Metastasis | interventions — Propranolol; tislelizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label interventional study evaluating the combination of propranolol, tislelizumab and GC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Propranolol + Tislelizumab + Gemcitabine/Cisplatin (Experimental): Patients will receive oral propranolol in combination with intravenous tislelizumab and gemcitabine/cisplatin as neoadjuvant therapy prior to radical surgery. Propranolol will be administered in escalating doses up to a maximum of 40 mg twice daily if tolerated. Tislelizumab is given intravenously every treatment cycle. Gemcitabine and cisplatin will be administered according to standard GC chemotherapy dosing. Participants will be monitored for treatment-related adverse events, including cardiovascular, hematologic, and immune-related toxicities. Dose adjustments, treatment interruptions, or discontinuation may be implemented according to predefined safety criteria.
  Interventions: Drug: propranolol; Drug: Tislelizumab; Drug: gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: propranolol — Propranolol will be administered orally as a non-selective β-adrenergic receptor blocker. Treatment will start at a low dose and may be escalated to a maximum of 40 mg twice daily if tolerated. Vital signs will be monitored regularly, and dose adjustment, interruption, or discontinuation may occur based on predefined cardiovascular safety criteria.
  Other Names: β-blocker; Propranolol Hydrochloride
Drug: Tislelizumab — Tislelizumab will be administered intravenously as an anti-PD-1 monoclonal antibody according to standard dosing schedules for neoadjuvant immunotherapy. Infusion monitoring will be conducted in a facility equipped for emergency management. Dose interruption or discontinuation may occur if immune-related adverse events develop.
Drug: gemcitabine — Gemcitabine will be administered intravenously as part of the gemcitabine/cisplatin chemotherapy regimen during neoadjuvant treatment. Hematologic parameters and organ function will be regularly monitored, and chemotherapy dose may be modified based on toxicity and tolerability according to institutional standards.
Drug: Cisplatin — Cisplatin will be administered intravenously as part of the gemcitabine/cisplatin regimen. Renal function, electrolyte balance, and hematologic tests will be routinely monitored. Dosing may be adjusted or withheld according to predefined safety criteria and institutional guidelines for cisplatin-based chemotherapy.

SUMMARY:
This is a prospective, multicenter, Phase Ib clinical study designed to evaluate the safety and preliminary efficacy of propranolol combined with tislelizumab plus gemcitabine/cisplatin (GC) as neoadjuvant therapy for patients with bladder urothelial carcinoma with clinical lymph node involvement (cT1-T4aN1-3M0). Current neoadjuvant immunochemotherapy regimens can improve clinical outcomes in cisplatin-eligible patients; however, patients with lymph node metastasis show a significantly poorer pathological complete response (pCR) rate compared with non-metastatic cases. Real-world clinical observations have shown that more than 20% of patients achieve complete response in the primary tumor after immunotherapy but have persistent or progressive positive lymph nodes, suggesting unique resistance mechanisms within lymph node metastatic lesions.

Preclinical studies conducted by our team demonstrated that sympathetic innervation within lymph nodes releases norepinephrine, which activates β-adrenergic signaling in metastatic tumor cells and promotes lipid metabolic reprogramming, leading to CD8⁺ T-cell exhaustion and immune resistance. Propranolol, a non-selective β-adrenergic blocker, may reduce metabolic stress and restore antitumor immunity, potentially enhancing the efficacy of immune checkpoint blockade.

In this study, enrolled patients will receive oral propranolol in combination with intravenous tislelizumab and standard GC chemotherapy prior to surgery. Participants will be closely monitored for treatment-related adverse events, including cardiovascular events, hematologic toxicity, and immune-related reactions. The primary endpoint is dose-limiting toxicity (DLT). Secondary endpoints include pathological complete response (pCR), pathological downstaging, safety, and survival outcomes. Exploratory analyses will evaluate changes in immune cell populations in tumor tissues, lymph nodes, and peripheral blood.

The results of this study aim to provide evidence for new neoadjuvant strategies targeting lymph node metastatic bladder cancer and support the development of personalized therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agrees to participate in the study, is able to provide written informed consent, and is willing to comply with study procedures and visit schedules.
2. Age ≥ 18 years at the time of consent; sex unrestricted.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
4. Histologically confirmed bladder urothelial carcinoma with clinical lymph node involvement (cT1-T4a, N1-N3, M0) based on the AJCC 8th edition. Mixed histology is permitted if the urothelial carcinoma component is ≥ 50%.
5. No antihypertensive medication used during screening, with resting systolic blood pressure between 110-140 mmHg measured under natural conditions.
6. Adequate organ function as demonstrated by laboratory results obtained within 14 days prior to enrollment:

   a. No administration of hematopoietic growth factors within 14 days prior to sample collection.

   i. Absolute neutrophil count ≥ 1.5 × 10⁹/L ii. Platelet count ≥ 90 × 10⁹/L iii. Hemoglobin ≥ 90 g/L b. INR or aPTT ≤ 1.5 × ULN c. Total bilirubin ≤ 1.5 × ULN (≤ 3 × ULN in patients with Gilbert syndrome or indirect hyperbilirubinemia) d. AST, ALT, and alkaline phosphatase ≤ 2.5 × ULN e. Preoperative pulmonary function assessment indicating tolerance of major abdominal surgery.
7. Cisplatin-eligible patients, or cisplatin-ineligible patients who meet at least one of the following:

   * ECOG performance status > 1 or Karnofsky 60-70%
   * Creatinine clearance < 60 mL/min
   * Grade ≥ 2 hearing loss (NCI-CTCAE v5.0)
   * Grade ≥ 2 peripheral neuropathy (NCI-CTCAE v5.0)
   * New York Heart Association (NYHA) class III or above heart failure
8. Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to enrollment and agree to use effective contraception during the study and for ≥ 120 days after the last dose. Male participants must agree to use effective contraception during the study and for ≥ 120 days after the last dose.

Exclusion Criteria:

1. Prior treatment with PD-1, PD-L1, PD-L2, CTLA-4 inhibitors, or other T-cell co-stimulatory/checkpoint agents.
2. Systemic antineoplastic therapy or immunomodulatory therapy within 28 days prior to enrollment, including interferon, interleukin-2, or TNF-based agents.
3. Prior radiotherapy for bladder cancer.
4. Prior systemic anticancer therapy except:

   1. Previous systemic chemotherapy completed ≥ 12 months before initiation of study treatment.
   2. Intravesical chemotherapy or immunotherapy completed ≥ 7 days prior to initiation of study treatment.
5. Major surgery or significant trauma within 28 days prior to enrollment (vascular access placement and TURBT excluded).
6. Receipt of live attenuated vaccines within 28 days prior to enrollment. Inactivated influenza vaccination is allowed; intranasal influenza vaccine is not permitted.
7. Active autoimmune disease requiring systemic therapy, as judged by the investigator.
8. Long-term systemic corticosteroid therapy or other immunosuppressive medications judged to interfere with study treatment.
9. Uncontrolled systemic disease that may interfere with treatment, including:

   * Clinically relevant electrolyte abnormalities
   * Hypoalbuminemia
   * Interstitial lung disease or non-infectious pneumonitis
   * Uncontrolled diabetes, hypertension, or cardiovascular disease (including unstable angina, myocardial infarction, symptomatic heart failure, or medically managed ventricular arrhythmias within 6 months).
10. Chronic hepatitis B infection with HBV DNA ≥ 500 IU/mL (2,500 copies/mL). Patients with inactive HBsAg carrier status or viral suppression (HBV DNA < 500 IU/mL) after antiviral therapy may be enrolled. HBV DNA testing is required if anti-HBc is positive.
11. Active hepatitis C infection. Patients who are HCV antibody negative, or HCV antibody positive but HCV RNA negative, are eligible.
12. History of immunodeficiency disorders (including HIV infection), congenital or acquired immune deficiency, or prior allogeneic stem cell transplantation or organ transplantation.
13. Known hypersensitivity to monoclonal antibodies, or known allergy to propranolol or other β-adrenergic receptor blockers.
14. Toxicities from previous therapies have not returned to baseline or stabilized, unless deemed not to pose a safety risk by the investigator (e.g., alopecia, neuropathy, specific laboratory abnormalities).
15. Contraindications to propranolol, including but not limited to:

    * Unstable angina
    * Decompensated heart failure
    * Symptomatic sinus bradycardia
    * Atrioventricular block
    * Severe asthma or bronchospasm
16. Current use of oral or intravenous β-blockers (e.g., atenolol, bisoprolol, carvedilol, metoprolol) that cannot be safely discontinued or transitioned. If previously used, a washout period of at least 14 days with medical reassessment is required before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) | At the end of Cycle 1 (each cycle is 28 days)
  Dose-limiting toxicities (DLTs) are defined as treatment-related adverse events occurring during the first treatment cycle that meet predefined severity criteria based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. DLTs may include grade 3 or higher non-hematologic toxicity, grade 4 hematologic toxicity, or clinically significant events leading to treatment interruption or discontinuation, as determined by the investigators.

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) Rate | At the time of surgery
  Pathological complete response (pCR) is defined as the absence of any residual tumor in the primary bladder lesion and in all examined regional lymph nodes following neoadjuvant therapy and surgical resection (pT0N0). The proportion of participants achieving pCR will be calculated relative to the total number of evaluable participants.
Pathological Downstaging Rate | At the time of surgery
  Pathological downstaging is defined as a postoperative pathological tumor stage (ypT) lower than the baseline clinical stage (cT), with downstaging to ypT2 or lower considered as treatment-induced downstaging. The proportion of evaluable participants achieving pathological downstaging will be recorded.
Incidence of Treatment-Related Adverse Events | From first dose through 30 days after the last administration of study treatment
  Adverse events (AEs), adverse drug reactions (ADRs), and serious adverse events (SAEs) will be collected and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Events will be summarized by frequency, severity grade, and relationship to study treatment.
Progression-Free Survival (PFS) | Up to 24 months after surgery
  PFS is defined as the time from study enrollment to the first documented disease progression, local or distant recurrence, or death from any cause, whichever occurs first. Participants without an event will be censored at the date of last disease assessment.
Overall Survival (OS) | Up to 36 months after surgery
  OS is defined as the time from study enrollment to death from any cause. Participants who remain alive at the end of follow-up will be censored at the date of last known contact.

OTHER OUTCOMES:
Proportion of exhausted CD8+ T cells among CD8+ T cells | At baseline and at time of surgery
  The proportion of exhausted CD8+ T cells (identified as PD-1⁺ TIM-3⁺ CD8⁺ cells) will be quantified in tumor tissue, lymph node samples, or peripheral blood mononuclear cells obtained before and after neoadjuvant treatment.